CLINICAL TRIAL: NCT05225909
Title: Multi-centre Prospective Observational Cohort Study: To Assess the Performance of Single Use Duodenoscope (aScope)
Brief Title: aScope Single Use ERCP Study- ASSURE Study
Acronym: ASSURE
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21GA088
Record Dates: First submitted 2022-01-21; First posted 2022-02-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: ERCP; Cholangitis; Infection
Keywords: aScope; Ambu Ltd
MeSH Terms: conditions — Cholangitis; Infections | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who Undergo ERCP procedure with aScope: This will be patients who undergo ERCP procedure using aScope.
  Interventions: Device: Endoscopic retrograde Cholangio-pancreatography (ERCP) with aScope (Single use duodenoscope

INTERVENTIONS:
Device: Endoscopic retrograde Cholangio-pancreatography (ERCP) with aScope (Single use duodenoscope — ERCP Procedure will be done using aScope. We will assess the performance of the aScope.

SUMMARY:
Patients undergo ERCP procedure (Endoscopic procedure with the help of x-rays) for a variety of reasons such as common bile duct (CBD)stones, bile duct obstruction secondary to bile duct narrowing (Strictures) and for bile leak. The incidence of infection post-ERCP is around one in 200. There are some group of patients where this risk is significantly increased. In this high risk group, the risk increases from 1 in 75 to in some diseases 1 in 15 (Described in PIS). There are some reports that some of the infection may be contributed by contamination of bacteria in the scope. This happens even after diligently sterilizing the scope. A multi-centre study reported that the risk of contamination is as high as 39% but what we do not know is how many resulted in bacterial infection. The investigators do not know what percentage of infection is secondary to the above. The new single use duodenoscope (aScope, Ambu Ltd) has been introduced in to the market to minimise the risk of post ERCP infection. It is CE marked but the evidence for performance of the aScope is limited. The investigators want to assess the performance of the scope simultaneously in multiple different hospitals. In addition, the investigators also want to assess the cost consequence to the NHS for using the above scope. Hence, the investigators want to assess the performance of the scope in the high risk groups for infection.

DETAILED DESCRIPTION:
ERCP is a therapeutic endoscopic procedure done to establish either bile duct or pancreatic duct drainage or both. The indications for ERCP are bile duct stones, bile duct strictures, sphincter of Oddi manometry with sphincterotomy, bile leak, pancreatic duct stones and pancreatic duct stricture. The intended benefits of the procedure are either to relieve bile duct/ pancreatic duct obstruction or facilitate bile duct/ pancreatic duct drainage. It is a minimally invasive procedure and is associated with reduced morbidity compared to surgery.

Gall stones are made of cholesterol, pigment and mixture of cholesterol and pigment. The incidence of stones with in the bile-duct varies from 4.6% to 19%.The stones are predominantly formed in the gall bladder and are displaced from the gall bladder in to the bile duct via the cystic duct. ERCP is an effective and minimally invasive treatment for bile duct stones. Treatment of extrahepatic biliary strictures; irrespective of their aetiology, is to place a stent across the stricture through ERCP and facilitate biliary drainage.

There is emerging data that the incidence of carbapenem resistant enterobacteriae, Multidrug-resistant Klebsiella pneumoniae, and New Delhi metallo-β-lactamase-producing carbapenem-resistant Escherichia coli (CRE) following exposure to contaminated duodenoscopes (ERCP endoscopes). The main reason for the outbreaks is due to inadequate reprocessing (Cleaning of endoscope post procedure) leading to contamination of endoscopes. To minimize the risk of contamination and outbreak of above infections, single use disposable duodenoscopes have been brought in to the market. The aim of the study is to assess the performance of the single use duodenoscope and the cost consequences associated with the above.

ELIGIBILITY:
Inclusion Criteria:

Patients who are at high risk of post ERCP infection such as

* Jaundice (Bilirubin >21)
* Primary sclerosing cholangitis
* Post liver transplant anastomotic stricture
* Inpatients
* Combined procedures (Ex: ERCP+ spy glass cholangioscopy)
* Previous inadequate biliary drainage.
* Biliary stricture
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Grade 1-3 ERCP on complexity grading (ASGE grading)
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

Patients with CBD stones and no jaundice

* Sphincter of Oddi manometry.
* Female participants who is pregnant, lactating or planning pregnancy during the course of the study.
* Patients who are unable to consent for the study.
* ERCP for Pancreatic pathology.
* Grade 4 complex ERCP (ASGE grading)
* Participant who is terminally ill /ECOG 4
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied will be patients who need ERCP procedure. All consecutive patients who are referred for ERCP will be screened to see if they meet the eligibility criteria to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Completion the intended ERCP procedure with single use duodenoscope. | 60-120 minutes
  To assess if the intended ERCP procedure can be successfully completed with single use disposable duodenoscope.

SECONDARY OUTCOMES:
Rate of complications | 30 days post procedure
  Complications associated with the procedure such as bleeding, pancreatitis, post-ERCP infection and perforation
Endoscopy metrics | 15 minutes after the procedure
  Endoscopy metric will be assessed through a agreed, structured questionnaire
Quality of life following the procedure | 5 minutes on day 7 and 30
  Quality of life will me measured using validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Suresh V Venkatachalapathy, MRCP, Study Chair — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
National research ethics committee does not allow sharing individual participant data because of confidentiality